CLINICAL TRIAL: NCT00583427
Title: Sulodexide Treatment in Patients With Dense Deposit Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: This study put on inactive status due to no identifiable subjects to enter the protocol.
Sponsor: University of Iowa (Other)
Responsible Party: Richard JH Smith, MD, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 200704758
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Dense Deposit Disease
MeSH Terms: conditions — Glomerulonephritis, Membranoproliferative | interventions — glucuronyl glucosamine glycan sulfate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sulodexide (Experimental)
  Interventions: Drug: Sulodexide

INTERVENTIONS:
Drug: Sulodexide — 200 mg per day in an oral gelcap form
  Other Names: KRX-101 (sulodexide)

SUMMARY:
The purpose of this study is to see if a medicine called Sulodexide will help prevent or slow down the progression of Membranoproliferative Glomerulonephritis type II/Dense Deposit Disease. Sulodexide is not yet FDA approved and has not been studied in children.

Study aim/hypotheses: to measure the efficacy of Sulodexide treatment in patients with the above disease/s.

DETAILED DESCRIPTION:
Study subjects will be asked to take Sulodexide twice a day. The Sulodexide will be taken in addition to the regular medications the subject is on. There will be no change in these other medications. The subject will also be asked to have blood tests each month to follow kidney function. The frequency of these tests is the normal/standard frequency for persons with MPGN II/DDD and is neither increased nor decreased because of participation in this study. The study will occur over 6 months for each subject.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 5 yrs. to 20 yrs. old
2. Patients must have Membranoproliferative Glomerulonephritis Type II (MPGN2), also known as Dense Deposit Disease (DDD)

Exclusion Criteria:

1. Patients less than 5 years of age or older than 20 years of age
2. Patients who DO NOT have a diagnosis of Membranoproliferative Glomerulonephritis (MPGN 2) also known as Dense Deposit Disease
3. Evidence of hepatic dysfunction including total bilirubin >2.0mg/dL (34 micromol/L) or liver enzymes >3 times upper limit of normal.
4. A history of any major medical condition (excluding DDD), including but not limited to: gastrointestinal bleeding in the past 3 months; HIV; active Hepatitis B or C (current active disease defined as an abnormal liver biopsy or persistent, elevated transaminases, SGOT, SGPT); and other medical conditions deemed serious by the investigator
5. any risk of bleeding, including a history of bleeding diathesis and a platelet count <100,000/mm3
6. active cancer
7. Participation in any experimental drug study in the 60 days prior to entry into this study; or plan to participate in any experimental drug study during the study period.
8. Known allergy or intolerance to any heparin-like compounds
9. Inability to give an informed consent or cooperate with the study personnel -

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2007-12; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
To see if Sulodexide will prevent or slow down the progression of DDD | 6 mo.

SECONDARY OUTCOMES:
Normalization of complement function | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Richard JH Smith, MD, Principal Investigator — University of Iowa
Locations (1):
- Richard Smith, MD, Iowa City, Iowa, United States